CLINICAL TRIAL: NCT06024031
Title: N-acetyl-L-cysteine for Promoting Hematopoietic Recovery in Patients With Acute Myeloid Leukemia After Chemotherapy--a Prospective Single-arm Clinical Study
Brief Title: NAC for Promoting Hematopoietic Recovery in Patients With Acute Myeloid Leukemia After Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAC for hematopoietic recovery
Record Dates: First submitted 2023-08-24; First posted 2023-09-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: From the first day after the end of chemotherapy: NAC 400mg tid D1-D28 was added on the basis of routine supportive therapy (blood transfusion)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAC group (Experimental): Low, intermediate risk AML patients were enrolled, and NAC (400mg tid) was administered orally from day1 to day 28 (D1-D28) after the end of induction chemotherapy.
  Interventions: Drug: N-acetyl-L-cysteine

INTERVENTIONS:
Drug: N-acetyl-L-cysteine — N-acetyl-L-cysteine (Yiweishi) capsules (Guangdong Renrenkang Pharmaceutical Industry) will be given orally 400mg three times a day from day 1 to day 28 after chemotherapy. In case of drug allergy such as nausea, vomiting, rash and bronchospasm, and disease relapse, to discontinue the drug immediately.
  Other Names: NAC (Yiweishi)

SUMMARY:
This is a prospective single-arm clinical study to evaluate the role of NAC after chemotherapy among patients with AML can promote hematopoietic recovery and does not affect the remission rate of the leukemia.

DETAILED DESCRIPTION:
Hematopoietic recovery after chemotherapy is an important factor affecting the prognosis of acute myeloid leukemia. A previous clinical prospective cohort study showed that NAC could improve the function of bone marrow endothelial progenitor cells after chemotherapy, without affecting leukemia cells. Previous animal models have found that chemotherapy can reverse the function of bone marrow endothelial cells in classic AML mice. NAC promotes hematopoietic recovery in AML mice by improving the bone marrow endothelial cells reversed by chemotherapy. Therefore, we hypothesized that the prophylactic administration of NAC after chemotherapy could facilitate the recovery of hematopoietic capacity by improving the bone marrow microenvironment of patients with AML.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed AML (except AML-M3)
2. Low-, intermediate risk AML (according to 2022 ELN)
3. Aged 18-60
4. No severe organ injury 1) Creatinine < 1.5mg/dl 2) Hemobilirubin ≤ 1.5 X ULN 3) AST and ALT ≤ 3.0 X ULN 4) Cardiac ejection index ≥ 50%
5. No uncontrolled active infections
6. Sign informed consent form, have the ability to comply with study and follow-up procedures

Exclusion Criteria:

1. Hypersensitivity to NAC
2. History of bronchial asthma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to hematopoietic recovery post chemotherapy | Participants will be followed for 2 months post induction chemotherapy
  Time to hematopoietic recovery (white blood cell > 1×10^9/L, platelet > 20 ×10^9/L), the dosages of G-CSF, red blood cell transfusion,platelet transfusion.

SECONDARY OUTCOMES:
complete remission rate | Participants will be followed for 1 year post induction chemotherapy
  Number of participants with complete remission will be calculated at 1-month post induction chemotherapy
relapse-free survival | Participants will be followed for 1 year post induction chemotherapy
  Number of participants with morphologic relapse will be calculated at one year post Number of participants with morphologic relapse will be calculated at one year post-HSCT
overall survival | Participants will be followed for 1 year post diagnosed
  Number of participants survived for 1 year post diagnosed will be calculated.
Adverse reactions | Participants will be closely observed for NAC-related toxicities during the NAC administration until 1-month post induction chemotherapy.
  Liver function, renal function, respiratory syndrom assessed by CTCAE v4.0 during oral administration of NAC.

OTHER OUTCOMES:
Endothelial progenitor cells | Participants will be followed for 1-month post induction chemothrapy
  Bone marrow microenvironment was evaluated before and after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Yuan Kong, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu LJ, Li CY, Xing T, Wang Y, Jiang Q, Jiang H, Wang J, Tang FF, Chang YJ, Zhang XH, Kong Y, Huang XJ. N-acetyl-L-cysteine promoted hematopoietic recovery in patients with acute myeloid leukemia after complete remission--A pilot study. Cancer Lett. 2025 Aug 10;625:217812. doi: 10.1016/j.canlet.2025.217812. Epub 2025 May 20. PMID 40403956